CLINICAL TRIAL: NCT04316156
Title: Hospital-home Linkage Short-term Rehabilitation Therapy Using Real-time Interactive Digital Healthcare System in Patients With Breast Cancer; Randomized Controlled Trial, Assessor Blinding, Multi-center Study
Brief Title: Real-time Interactive Digital Healthcare System in Patients With Breast Cancer; Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SMC-2019-05-021 (2)
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Range of motion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise using Uincare Homeplus (Experimental): Uincare Homeplus
  Interventions: Device: Uincare Homeplus
- Exercise using brochure (Active Comparator): brochure
  Interventions: Other: Brochure

INTERVENTIONS:
Device: Uincare Homeplus — Interactive digital healthcare system
  Other Names: digital healthcare
  Arms: Exercise using Uincare Homeplus
Other: Brochure — Brochure
  Arms: Exercise using brochure

SUMMARY:
This study aims to examine the effect of hospital-home linkage short-term rehabilitation therapy using real-time interactive digital healthcare system (Uincare Homeplus) in post-operative patients with breast cancer. This is prospective study. 100 breast cancer patients who underwent axillary lymph node diessection or breast reconstruction following mastectomy will be examined, and those with limited range of motion (ROM) of affected shoulder will be enrolled in the study. Shoulder ROM, Quick-DASH, pain evaluation with NRS, quality of life evaluation with FACT-B and EQ-5D will be evaluated on enrollment, 4-week, 8-week, and 12-weeks after enrollment.

DETAILED DESCRIPTION:
The limited range of motion (ROM) of the shoulder occur often after receiving breast cancer surgery, which may be due to post-operative pain, stiffness of shoulder girdle muscle, and etc. Due to this limited ROM, the patients may have difficulty with activities of daily life and quality of life may be reduced.

Uincare Homeplus is software manufactured in Korea, which uses infrared, kinect camera and motion capture technology to track 3D motion of the patients' articulation. Using this technology, the patients can receive feedback of their motion immediately.

The objective of the study is to examine the effect of hospital-home linkage short-term rehabilitation therapy using real-time interactive digital healthcare system (Uincare Homeplus) in post-operative patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent breast cancer surgery (axillary lymph node dissection or breast reconstruction following mastectomy)
* Limited active/passive range of motion of the affected shoulder (Flexion <160' or Abduction <160')
* post-operative day not exceeding 8 week
* Patients who agreed informed consent

Exclusion Criteria:

* Bilateral breast cancer surgery
* Patients with shoulder pain and limited ROM before breast cancer surgery
* Those unable to perform exercise due to general deconditioning
* Those with communication difficulty

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Range of motion in affected shoulder | Enrollment, 4 week, 8 week, 12 week
  Evaluation of change in range of motion of the affected shoulder from baseline to 12 weeks

SECONDARY OUTCOMES:
Numerical rating scale of affected shoulder | Enrollment, 4 week, 8 week, 12 week
  Evaluation of pain in the affected shoulder using numerical rating scale minimum ~ maximum value: 0 ~ 10, higher scores mean worse outcome.
Functional outcome (Quick Disability of Arm, Shoulder, Hand) | Enrollment, 4 week, 8 week, 12 week
  Evaluation of shoulder function using Quick Disability of Arm, Shoulder, Hand (Quick DASH) ranging from 0 (no disability) to 100 (most severe disability).
Quality of life in the patient with breast cancer (1) | Enrollment, 4 week, 8 week, 12 week
  Evaluation of quality of life using Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) The total FACT-B score ranges from 0 to 123, and is calculated by adding the scores from each of these subscales. Lower scores indicate better health.
Quality of life in the patient with breast cancer (2) | Enrollment, 4 week, 8 week, 12 week
  Evaluation of quality of life using EQ-5D-5L. This scale is numbered from -0.066 to 0.904. lower value means the worst quality of life you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: JIHYE HWANG, Professor, Study Chair — Physical & Rehabilitation Medicine Samsung Medical Center
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Department of rehabilitation, Seoul St. Mary's Hospital, College of Medicine, The Catholic University of Korea, Seoul, Seocho-gu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park HY, Nam KE, Lim JY, Yeo SM, Lee JI, Hwang JH. Real-Time Interactive Digital Health Care System for Postoperative Breast Cancer Patients: A Randomized Controlled Trial. Telemed J E Health. 2023 Jul;29(7):1057-1067. doi: 10.1089/tmj.2022.0360. Epub 2022 Nov 29. PMID 36454316
- [Derived] Park HY, Nam KE, Lim JY, Yeo SM, In Lee J, Hwang JH. Real-time interactive digital healthcare system for post-operative breast cancer patients: study protocol for a randomized controlled trial. Trials. 2021 Aug 19;22(1):549. doi: 10.1186/s13063-021-05535-8. PMID 34412658